CLINICAL TRIAL: NCT03740802
Title: Evaluation of Hypophosphatemia as a Predictor of Sepsis in Surgical Resuscitation Units.
Brief Title: Hypophosphatemia as a Predictor in Surgical Resuscitation Sepsis
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PORPOISE2-REA (29BRC18.0022)
Record Dates: First submitted 2018-04-25; First posted 2018-11-14 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-01

CONDITIONS: Hypophosphatemia; Infection
MeSH Terms: conditions — Hypophosphatemia; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective study in the surgical intensive care unit of the Brest Teaching Hospital (France) during a 6-months period (January 2015 -May 2015) to study the independent association between hypophosphatemia and 28-day infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults

Exclusion Criteria:

* Less than 18 years old
* Infected at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to 15-bed surgical ICU between January 1, 2015 and June 31, 2015 were screened for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with sepsis within 28 days after ICU admission | 28 days since the ICU admission
  Sepsis was defined according to the criteria of the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France